CLINICAL TRIAL: NCT00005866
Title: A Phase III Randomized Study Comparing Busulfan-Total Body Irradiation Versus Cyclophosphamide-Total Body Irradiation Preparative Regimen in Patients With Advanced Myelodysplastic Syndrome (MDS) or MDS-Related Acute Myeloid Leukemia (AML) Undergoing HLA-Identical Sibling Peripheral Blood Stem Cell Transplantation, (A BMT Study)
Brief Title: S9920 Busulfan Compared With Cyclophosphamide in Patients Undergoing Total-Body Irradiation Plus Peripheral Stem Cell Transplantation for Advanced Myelodysplastic Syndrome or Related Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S9920; S9920 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2004-03-16 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: untreated adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate; Radiotherapy

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: methotrexate; Procedure: allogeneic bone marrow transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: busulfan — arm 1: 0.44 mg/kg every 6 hours, IV over 2 hours, day -7 to -4
Drug: cyclophosphamide — arm 2: 60 mg/kg every 24 hrs for 2 doses, IV over 2 hrs, days -5 and -4
Drug: cyclosporine — both arms per published schedule
Drug: methotrexate — GVHD: 15 mg/m2 day 1, 10 mg/m2 day 3, 6 and 11 by IV
Procedure: allogeneic bone marrow transplantation — day 0
Radiation: radiation therapy — both arms: 1200 cGy total dose (6 x 200 fractions)

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells. It is not yet known if total-body irradiation plus peripheral stem cell transplantation is more effective with busulfan or with cyclophosphamide for myelodysplastic syndrome or acute myeloid leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of busulfan with that of cyclophosphamide in patients undergoing total-body irradiation plus peripheral stem cell transplantation for advanced myelodysplastic syndrome or related acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare event free survival after total body irradiation (TBI) plus busulfan versus TBI plus cyclophosphamide followed by allogeneic peripheral blood stem cell transplantation in patients with advanced myelodysplastic syndrome (MDS) or MDS related acute myeloid leukemia. II. Determine the distribution of pharmacokinetic parameters for busulfan in those patients randomized to the busulfan treatment arm. III. Investigate the prognostic significance for event free survival of prior history of red cell transfusions, cytogenetic pattern, and of functional drug resistance at diagnosis in these patients. IV. Estimate the frequencies of cytogenetic and genetic changes during disease progression in these patients.

OUTLINE: This a randomized, multicenter study. Patients are stratified according to age (40 and under vs 41-55) and diagnosis and International Prognostic Scoring System (IPSS) risk group (myelodysplastic syndrome (MDS)/IPSS - intermediate 1 vs MDS/IPSS - intermediate 2 vs MDS/IPSS high risk vs MDS related acute myeloid leukemia). Patients are randomized to one of two treatment arms. Arm I: Patients receive busulfan IV over 2 hours every 6 hours on days -7 to -4 for a total of 16 doses. Arm II: Patients receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients receive total body irradiation (TBI) twice a day on days -3 to -1; peripheral blood stem cell transplantation from genotypically HLA identical sibling on day 0; cyclosporine IV every 12 hours on days -1 to 60, and then tapering in the absence of graft versus host disease; and methotrexate IV on days 1, 3, 6, and 11. Patients are followed every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 240 patients (120 per treatment arm) will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytologically confirmed myelodysplastic syndrome (MDS) Increased blasts (i.e., greater than 1 to 30% peripheral blood blasts and/or 5 to 30% bone marrow blasts) AND International Prognostic Score intermediate 1, intermediate 2, or high risk Refractory anemia with excess blasts OR Refractory anemia with excess blasts in transformation (no presence of auer rods as sole criteria) OR Chronic myelomonocytic leukemia Greater than 1% blasts in the peripheral blood and/or at least 5% blasts in the bone marrow OR MDS related acute myeloid leukemia Arising after documented MDS of at least 60 days Absolute peripheral blast count no greater than 5,000/mm3 Must have genotypically HLA identical sibling donor Must also be enrolled on SWOG-S9910 and SWOG-9007

PATIENT CHARACTERISTICS: Age: 16 to 55 Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified Other: No prior malignancy within past 5 years except: Adequately treated basal cell or squamous cell skin cancer Carcinoma in situ of the cervix Adequately treated stage I or II cancer in complete remission HIV negative Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No autologous peripheral stem cell transplantation prior to diagnosis of myelodysplastic syndrome (MDS) or MDS related acute myeloid leukemia Chemotherapy: No prior chemotherapy for MDS or MDS related acute myeloid leukemia except oral chemotherapy to control leukocytosis or thrombocytosis (e.g., hydroxyurea or etoposide) Endocrine therapy: Not specified Radiotherapy: No radiotherapy prior to diagnosis of MDS or MDS related acute myeloid leukemia Surgery: Not specified

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2000-02; Primary Completion 2004-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival | every 6 months after stem cell infusion until death or 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne E. Anderson, MD, Study Chair — Katmai Oncology Group
Locations (66):
- United States (65):
  - Good Samaritan Medical Center, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Scripps Clinic, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - St. Joseph Hospital - Orange, Orange, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - Northern California Cancer Specialists Medical Clinic, Walnut Creek, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Memorial Medical Center, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Cancer Research Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. John's Health System, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Jewish Hospital of Cincinnati, Inc., Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Legacy Cancer Services, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - Health Science Center, Lubbock, Texas
  - Methodist Health Care System, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Franciscan Health System, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
- Princess Margaret Hospital, Toronto, Ontario, Canada